CLINICAL TRIAL: NCT06037642
Title: All Children in Focus (ABC) 0-2 Years: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Anders Kassman, Associate professor, Ersta Sköndal University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: All children in focus
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Parent-Child Relations; Parenting
Keywords: Parenting support
MeSH Terms: interventions — abacavir; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: ABC 0-2 years
- Control group (Active Comparator)
  Interventions: Other: waiting list

INTERVENTIONS:
Behavioral: ABC 0-2 years — Four 1 hour meetings and homework
  Arms: Intervention group
Other: waiting list — Will be put on hold for four weeks
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare parents tools to handle challenges and strengths as parents. The main questions it aims to answer are:

* Do participating parents feel more confident than non partipating parents?
* Does the program have positive effects on parenting practices, parents´ well-being, and social support?
* Is the programme more effective for some groups of parents ( e.g., gender, socioeconomis status)

Participating parents will attend four 1-hour, manual based sessions followed by a 30-minutes optional coffe break. In addition parents will be asked to do homework assignments between the sessions.

Researchers will compare the intervention group with an equally sized control group that will receive the program later the same year.

ELIGIBILITY:
Inclusion Criteria:

Parents to children aged 0-2 years

Exclusion Criteria:

Non fluent in Swedish language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Parents´self efficacy | Four weeks
  Questionnaire
Parenting practices and parent child relationship | Four weeks
  Questionnaire
Parents´involvement and warmth | Four weeks
  Questionnaire
Parents´ well-being | Four weeks
  Questionnaire
Parents´ social network | Four weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Eriksson, Phd, Study Director — Ersta Sköndal University College
Locations (1):
- PLUS, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No